CLINICAL TRIAL: NCT03883750
Title: Induced Pluripotent Stem Cells for the Development of Novel Drug Therapies for Hepatic and Neurological Niemann Pick Disease
Brief Title: Induced Pluripotent Stem Cells for Niemann Pick Disease
Acronym: IPSNPABC
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: IPSNPABC 6-2018
Record Dates: First submitted 2019-03-04; First posted 2019-03-21 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2020-04

CONDITIONS: Niemann-Pick Diseases
MeSH Terms: conditions — Niemann-Pick Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The skin biopsy will be carried out for patients with a diagnosis of Niemann Pick. The biopsy is performed by the physician by means of punch biopsy (diameter 2-3 mm) under local anesthesia, preferably on the forearm (alternatively: thigh). The biopsy is immediately transferred to sterile cell culture medium and sent by center representative for the quickest possible processing to CENTOGENE's laboratory located in Germany or to professional collaborators being part of the project.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Establishment of individualized human cellular disease models based on induced pluripotent stem cells that reflect the broad heterogeneous phenotypic spectrum of Niemann Pick disease

DETAILED DESCRIPTION:
Niemann-Pick disease type C (NPC) is a lipid storage disease that can present in infants, children, or adults. Neonates can present with ascites and severe liver disease from infiltration of the liver and/or respiratory failure from infiltration of the lungs. Other infants, without liver or pulmonary disease, have hypotonia and developmental delay. The classic presentation occurs in mid-to-late childhood with the insidious onset of ataxia, vertical supranuclear gaze palsy, and dementia. Dystonia and seizures are common. Dysarthria and dysphagia eventually become disabling, making oral feeding impossible; death usually occurs in the late second or third decade from aspiration pneumonia. Adults are more likely to present with dementia or psychiatric symptoms. The diagnosis of NPC is confirmed by biochemical testing that demonstrates impaired cholesterol esterification and positive filipin staining in cultured fibroblasts. Biochemical testing for carrier status is unreliable. Most individuals with NPC have NPC1, caused by mutations in the NPC1 gene; fewer than 20 individuals have been diagnosed with NPC2, caused by mutations in the NPC2 gene. Molecular genetic testing of the NPC1 genes detects disease-causing mutations in approximately 94% of individuals with NPC. Such testing is available clinically.

NPC is inherited in an autosomal recessive manner. The phenotype (i.e., age of onset and severity of symptoms) usually runs true in families. Carrier testing for at-risk relatives and prenatal testing for pregnancies at increased risk are possible when the two disease-causing mutations have been identified in the family.

Though NPC is a pan-ethnic disorder, the prevalence of this autosomal-recessive disorder is elevated in countries with a higher frequency of consanguinity.

Therefore, the goal of the study to prepare a cell culture from patients affected with Niemann Pick disease in order to identify novel pathways and proteins involved in disease progression that allow for an earlier diagnosis (i.e. before symptom onset) and that are suitable targets for an individualized therapeutic approach able to address not only the hepatic form, but also the neurologic form of the disease, which is less responsive to the current therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained from the patient or the parents before any study related procedures
* Patients of both genders older than 6 months and younger than 80 years
* The patient has a diagnosis of Niemann Pick disease

Exclusion Criteria:

* No Informed consent from the patient or the parents before any study related procedures
* Patients of both genders younger than 6 months or older than 80 years
* No diagnosis of Niemann Pick disease

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient has a diagnosis of Niemann Pick disease
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
To generate patient-specific induced pluripotent stem cells and then differentiate them into neural cells | 24 months
  The aim of this study is to generate patient-specific induced pluripotent stem cells and then differentiate them into neural cells to study the misfolded proteins in endoplasmic reticulum, their role in untranslated protein response, and possible mechanisms to shuttle the misfolded proteins into lysosomes.

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Rolfs, Prof., Principal Investigator — CENTOGENE GmbH Rostock
Locations (1):
- Childrens Hospital and Institute of Child Health, Ferozepur Road, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided